CLINICAL TRIAL: NCT04369417
Title: Evaluation of a Resiliency Intervention for Siblings of Children With Autism Spectrum Disorder (ASD)
Acronym: SibChat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Karen Kuhlthau, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2019P003218
Record Dates: First submitted 2020-02-20; First posted 2020-04-30 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Stress
Keywords: Resiliency Training; Autism Spectrum Disorder; Family Relationships
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: 3RP treatment (Experimental): An adapted version of the Relaxation Response Resiliency Program (3RP) for siblings of children with ASD. The adapted program incorporates the three prongs of the 3RP: RR elicitation, stress awareness, and adaptive strategies.
  Interventions: Behavioral: Relaxation Response Resiliency Program for Siblings of Children with ASD
- Active Comparator: Waitlist control (Active Comparator): An adapted version of the Relaxation Response Resiliency Program (3RP) for siblings of children with ASD. The adapted program incorporates the three prongs of the 3RP: RR elicitation, stress awareness, and adaptive strategies.
  Interventions: Behavioral: Relaxation Response Resiliency Program for Siblings of Children with ASD

INTERVENTIONS:
Behavioral: Relaxation Response Resiliency Program for Siblings of Children with ASD — Virtually delivered psycho-educational resiliency training program for teenage siblings of children with ASD.

SUMMARY:
The proposed research has the following objectives:

Based off findings from the "Development of a Resiliency Program for Siblings of Children with Autism Spectrum Disorder" qualitative focus group study (protocol 2019P002284), the aim is to determine the feasibility and acceptability, of an 8-session Relaxation Response Resiliency (SibChat) program for siblings of children with ASD.

We primarily aim to test the preliminary effectiveness of a pilot waitlist controlled trial on improving resiliency and stress coping, This will be assessed by comparing Baseline-3 mo. scores on primary and secondary outcome measures between the Immediate and Waitlist control groups.

Among participants randomized to both conditions, we secondarily aim to investigate the extent of pre-post changes in primary and secondary outcomes. Among immediate condition group only, we also aim to assess whether end-of-treatment (3 mo. post enrollment) improvements will be sustained at 6-mo. post enrollment.

DETAILED DESCRIPTION:
This intervention will be a modified version of Dr. Elyse Park's evidence-based 8-week multimodal treatment which is designed to promote adaptation to stress and promotion of resiliency. The program is an 8 session, 1 hour a week multi modal intervention that incorporates relaxation techniques, stress awareness discussion, and adaptive strategies for coping with stress. This study will refine an 8-session group virtual-delivered resiliency treatment program consisting of 8 virtual group 1-1 ½ hour sessions. The goal of this study would be to advance our ultimate objective to implement a national sibling resiliency program.

ELIGIBILITY:
Inclusion Criteria:

1. Age 14-17 years (inclusive of ages 14 and 17)
2. Being the sibling of at least one individual with ASD
3. Access to internet or smart phone
4. English speaking

Exclusion Criteria:

1. Diagnosis of ASD
2. Past year psychiatric hospitalization

There are no exclusion criteria with respect to ethnicity or socioeconomic status.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Feasibility assessed by the number participants enrolled. | 6 months
  We will assess study feasibility based on number of participants enrolled in the study (target N=40)
Feasibility assessed by the number SibChat-3RP of sessions attended | 8 weeks
  Whether youth attended at least 5 out of 8 total program sessions.
Feasibility assessed by the survey retention post intervention. | 6 months
  Among participants randomized to both conditions, feasibility is assessed by the number of participants who completed the T2 and T3 surveys, 3 months and 6 months post baseline, respectively.
Acceptability assessed using the participant feedback survey | 3 months
  The participant feedback survey is a questionnaire made up of likert scales and open ended questions designed to record acceptability of the SibChat-3RP program on topics including length of sessions, number of sessions, and virtual delivery.
Acceptability assessed by relaxation response adherence | 3 months
  Among participants randomized to both conditions, relaxation response adherence is measured at T1, T2 and T3. Relaxation response adherence is a 1-item likert scale that indicates how often participants practice relaxation response exercises. Acceptability is determined based on whether participants indicate that they practice relaxation response exercises at least bimonthly 3 months post intervention.
Effectiveness of trial on improving stress coping ability (assessed using Measure of Current Status-A) | 3 months
  Measure of Current Status-A is a questionnaire - the score on the questionnaire is used to indicate stress coping ability. A change in score indicates a change in indicated stress coping ability. Comparison of intervention and wait list control 3 months after baseline (T1).
Effectiveness of trial on improving resiliency (assessed using Current Experiences Scale) | 3 months
  Current experiences Scale is a questionnaire. Improved resiliency is measured base upon change in questionnaire score. Comparison of intervention and wait list control 3 months after baseline (T1).

SECONDARY OUTCOMES:
Pre-post intervention changes as measured by change in primary outcome scores of resiliency and stress coping. | 3 months
  Among participants randomized to both conditions, pre-post intervention changes in primary outcome scores of resiliency and stress coping will be assessed using the scores from the questionnaire (includes all primary outcome scores indicated above).
Sustained improvements in primary outcomes of resiliency and stress coping as measured by sustained change in primary outcome scores. | 3 months
  Among immediate condition group only, assess whether end-of-treatment (3 mo. post enrollment) improvements in primary outcome scores (resiliency and stress coping indicated above; collected using a questionnaire) will be sustained at 6-mo. post enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Karen A Kuhlthau, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuhlthau KA, Traeger L, Luberto CM, Perez GK, Goshe BM, Fell L, Iannuzzi D, Park ER. Resiliency Intervention for Siblings of Children With Autism Spectrum Disorder: A Randomized Pilot Trial. Acad Pediatr. 2023 Aug;23(6):1187-1195. doi: 10.1016/j.acap.2022.11.011. Epub 2022 Nov 30. PMID 36460184